CLINICAL TRIAL: NCT01772836
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Ascending Single and Multiple-Dose Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Intravenous Biapenem (RPX2003) and RPX7009 Given Alone and in Combination in Healthy Adult Subjects.
Brief Title: Safety Study of Intravenous Biapenem (RPX2003) and RPX7009 Given Alone and in Combination
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rempex Pharmaceuticals (a wholly owned subsidiary of The Medicines Company) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Rempex 403
Record Dates: First submitted 2013-01-16; First posted 2013-01-21 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Healthy Volunteers; Bacterial Infections
MeSH Terms: conditions — Bacterial Infections | interventions — RPX7009; beta-Lactamase Inhibitors; biapenem; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Normal saline (Placebo Comparator): Single and multiple dose of normal saline
  Interventions: Drug: Normal saline
- Single dose IV of biapenem or RPX7009 (Experimental): Single dose IV infusion of biapenem or RPX7009
  Interventions: Drug: RPX7009; Drug: Biapenem
- Single dose of biapenem or RPX7009 (Experimental): Single IV dose of biapenem or RPX7009 (for those on active drug, this will be the drug not given in the first IV treatment)
  Interventions: Drug: RPX7009; Drug: Biapenem
- Biapenem and RPX7009 in combination (Experimental): Single dose followed by a multiple dose of biapenem and RPX7009 in combination
  Interventions: Drug: RPX7009; Drug: Biapenem

INTERVENTIONS:
Drug: RPX7009 — Up to three (3) cohorts of 10 healthy adult subjects (8 active, 2 placebo)
  Other Names: (beta-lactamase inhibitor)
  Arms: Biapenem and RPX7009 in combination; Single dose IV of biapenem or RPX7009; Single dose of biapenem or RPX7009
Drug: Biapenem — Up to three (3) cohorts of 10 healthy adult subjects (8 active, 2 placebo)
  Other Names: RPX2003
  Arms: Biapenem and RPX7009 in combination; Single dose IV of biapenem or RPX7009; Single dose of biapenem or RPX7009
Drug: Normal saline — Up to three (3) cohorts of 10 healthy adult subjects (8 active, 2 placebo)
  Other Names: Placebo
  Arms: Normal saline

SUMMARY:
RPX7009 (beta-lactamase inhibitor) is being studies in combination with a carbapenem biapenem to treat bacterial infections, including those due to multi-drug resistant bacteria.

DETAILED DESCRIPTION:
The worldwide spread of resistance to antibiotics among Gram-negative bacteria, particularly members of the ESKAPE group of pathogens, has resulted in a crisis in the treatment of hospital acquired infections. In particular, the recent dissemination of a serine carbapenemase (e.g., KPC) in Enterobacteriaceae in US hospitals now poses a considerable threat to the carbapenems and other members of the beta-lactam class of antimicrobial agents.

Rempex is developing a fixed combination antibiotic of a carbapenem (RPX2003 or biapenem) plus a new beta-lactamase inhibitor (RPX7009) which has activity against serine beta-lactamases, including KPC. This Phase 1 study will assess the safety, tolerability and pharmacokinetics and pharmacodynamics of Intravenous Biapenem and RPX7009, administered alone and in combination in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males and/or females, 18 to 55 years of age
* Body mass index (BMI) ≥ 18.5 and ≤ 29.9 (kg/m2) and weight between 55.0 and 100.0 kg (inclusive).
* Medically healthy with clinically insignificant screening results
* Non-tobacco/nicotine-containing product users for a minimum of 6 months prior to Day 1.
* Sexually abstinent or use acceptable methods of birth control

Exclusion Criteria:

* History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, or psychiatric disease.
* History or presence of alcoholism or drug abuse within the 2 years prior to Day 1.
* Hypersensitivity or idiosyncratic reaction to beta-lactam antibiotics (e.g. penicillins, cephalosporins, carbapenems, etc.).
* Use of any over-the-counter (OTC) medication, including herbal products and vitamins, within the 7 days prior to Day 1. Up to 2 grams per day of acetaminophen is allowed for acute events at the discretion of the PI.
* Plasma donation within 7 days prior to Day 1.
* Subjects who have any abnormalities on laboratory values at screening or check-in (Day -1).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Safety from baseline to the end of the study | Day 1 - Day 17
  Number of patients with adverse events; assessed by patient reporting, collection of vital signs, ECGs and absolute values and changes over time of hematology, chemistry and urinalysis.

SECONDARY OUTCOMES:
Composite of Pharmacokinetic (PK) parameters of RPX7009, biapenem & the combination following ascending single and multiple dose administration. | Day 1 - Day 14
  Comparison will be performed between the cohorts for the plasma AUC0-t, AUC0-inf, Cmax, and Tmax.
  Urine PK parameters such as amount excreted and % dose excreted will be calculated from urinary excretion data.
Composite of Pharmacodynamic (PD) parameters of RPX7009, biapenem & the combination following ascending single and multiple dose administration. | Days 1-14
  Serum for bactericidal titers (SBT) assessments will be collected on Days 1, 4, 7 and 14 (at the end-of-infusion (EOI)), and at 2, 4, and 8 hours after start of infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Jefferey Loutit, MBChB, Study Director — Sponsor GmbH
Locations (1):
- CMAX, Adelaide, South Australia, Australia